CLINICAL TRIAL: NCT02710825
Title: Single Center Randomized Clinical Trial, That Evaluates the Effect of Osteopathic Care on Postoperative Pain in Children With Congenital Heart Disease Surgery
Brief Title: Osteopathy and Children With Congenital Heart Disease Surgery
Acronym: OSCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Necker-Enfants Malades (Other)
Collaborators: ARCFA : Association for research in cardiology foetal to adult (Unknown)
Responsible Party: Principal Investigator, Marion Hery, Osteopath, Hôpital Necker-Enfants Malades
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-A01332-47
Record Dates: First submitted 2016-03-02; First posted 2016-03-17 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Osteopathic Physicians

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteopathic treatment (Experimental)
  Interventions: Other: Osteopathy
- Simulated osteopathic treatment (Placebo Comparator)
  Interventions: Other: superficial palpatory agreement

INTERVENTIONS:
Other: Osteopathy — The treatment begins, if possible, on the body part of the child whose osteopathic score is the highest , with the least elasticity and mobility. Then the other restricted joints will be treated. The set of techniques will be carried out after palpation and appropriate tensioning. The various actions will be carried out on the tissues and joints who have been particularly affected by the operation.
  When a joint or tissue has a restricted mobility in a direction or a specific movement, it will require appropriate and gently manual correction, in order to reduce and improve its functionality.
  Arms: Osteopathic treatment
Other: superficial palpatory agreement — The simulated treatment also begins with the body part of the child whose osteopathic score is the highest. Then the other restricted joints will be treated. The set of techniques will be carried out with the same investments as the tests , with a superficial palpatory agreement and without tensioning so that the restricted articulation or tissue will not be corrected
  Arms: Simulated osteopathic treatment

SUMMARY:
Osteopathic care impact on postoperative pain assessed by osteopathic session, evaluated by EVENDOL scale surgery on children with congenital heart disease

DETAILED DESCRIPTION:
The management of pain in children after cardiac surgery is the key to ensure a better comfort and fast home return.

Aside drugs and psychology or physical therapy, no other alternative is proposed in the medico-surgical unit of pediatric cardiology at the Necker hospital.

Following a feasibility study within the department, osteopathic care showed significant pain reduction in postoperative surgery assessed through the EVENDOL scale.

The goal was mainly to improve mobility restricted areas due to the operation, and so help to reduce post-operative pain.

Investigators propose to continue the assessment of the overall osteopathic taking care of the child after heart surgery while retaining EVENDOL scale as primary endpoint. Population will include children from the age of 5 days to less than 7 years old.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5 days to 7 years old
* Congenital heart sternotomy or thoracotomy operated
* Postoperative management at the Necker hospital in Paris, followed by Professor Damien Bonnet team
* Agreeing to participate of one of the holders of parental authority
* Oral Agreement child age
* Minimal knowledge of French language by parents
* Covered by the French social security system

Exclusion Criteria:

* Heart disease treated by interventional catheterization
* Postoperative complications requiring more than three weeks of intensive care
* Participation in an other biomedical research protocol
* Refusal or linguistic or mental disabilities or parents of the child

Ages: 5 Days to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Change of EVENDOL from day1 at day2 | day 2
  Pain Rating Scale and discomfort in children, giving a score from 0 to 15 filled by doctor

SECONDARY OUTCOMES:
Change of EVENDOL from day1 at day2 | day 2
  Pain Rating Scale and discomfort in children, giving a score from 0 to 15 filled by children's parent (mother or father)
Change of Score OSCAR from day1 at day2 OS : for osteopathy CAR : for cardiopathy | day 2
  Osteopathic Scale assessing the mobility of each part of the body to give a final score OSCAR ranging from 0 to 45.
Change of Faces scale or Visual analog scale from day1 at day2 | day 2
  Pain Rating Scale and discomfort in children giving a score from 0 to 10 filled by child
Change of Arterial Pressure from day1 at day2 | Day 2
Change of Oxygen saturation from day1 at day2 | day2
Change of cardiac frequency from day1 at day2 | day 2
Change of cardiac breathing frequency from day1 at day2 | day2
Analgesic intake at day1 | day1
  Doctor's drugs prescription
Analgesic intake at day2 | day2
  Doctor's drugs prescription

CONTACTS AND LOCATIONS:
Overall Officials: Fanny Bajolle, Ph, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hospital Necker, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guiney PA, Chou R, Vianna A, Lovenheim J. Effects of osteopathic manipulative treatment on pediatric patients with asthma: a randomized controlled trial. J Am Osteopath Assoc. 2005 Jan;105(1):7-12. PMID 15710659
- [Background] Degenhardt BF, Kuchera ML. Osteopathic evaluation and manipulative treatment in reducing the morbidity of otitis media: a pilot study. J Am Osteopath Assoc. 2006 Jun;106(6):327-34. PMID 16790538